CLINICAL TRIAL: NCT05130320
Title: SHINE: Severe Asthma Covid Vaccine Response Study
Brief Title: Severe Asthma Covid Vaccine Response Study
Acronym: SHINE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Asthma Allergy & Inflammation Research Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: RHM MED1777
Record Dates: First submitted 2021-05-07; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Coronavirus Antibody Levels

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Asthma biologics: 120 people receiving asthma biologics (monoclonal antibodies)
  Interventions: Other: Not Interventional their treatments are their routine NHS care
- Asthma inhalers: 40 people receiving asthma inhalers
  Interventions: Other: Not Interventional their treatments are their routine NHS care
- Steroid tablets: 40 people needing daily steroid tablets to control their asthma
  Interventions: Other: Not Interventional their treatments are their routine NHS care
- Healthy Control: 50 age-matched healthy people
  Interventions: Other: Not Interventional their treatments are their routine NHS care

INTERVENTIONS:
Other: Not Interventional their treatments are their routine NHS care — Not Interventional their treatments are their routine NHS care

SUMMARY:
This study aims to employ a simple finger-prick home test to detect post vaccination antibody levels. The investigators will compare antibody responses in patients with severe asthma on varying treatment regimes (biologics, daily steroids, inhalers-only) with healthy, age-matched controls to study if the magnitude and range of responses vary between severe asthmatics and healthy individuals.

DETAILED DESCRIPTION:
SARS-CoV-2 and the resulting COVID-19 pandemic has had a major impact on quality of life in people with severe asthma. Careful isolation and lockdown measures have protected many patients, but with major impacts on wellbeing and mental health. Vaccination opens a "light at the end of the tunnel" by protecting against COVID-19. However, the following questions remain unanswered for Covid vaccination in severe asthma: 1) What are patients' expectations/attitudes towards vaccination? 2) Will vaccines induce good immune responses which protect from Covid-19 infections? The first question is being addressed by a survey created SHARP, a European Clinical Research Collaboration on severe asthma- people with asthma from the UK and Europe will be invited to complete the survey. To complement this, the investigators propose a UK pilot study (carried out in up to four severe asthma centres) to measure immune responses following vaccination in 200 people with severe asthma. The investigators will invite 120 people receiving asthma biologics (monoclonal antibodies), 40 people receiving asthma inhalers, 40 people needing daily steroid tablets to control their asthma, and 50 age-matched healthy people. Immune responses will be studied using a simple home blood antibody test posted to participants. By pricking their finger, patients will collect 5-6 drops of blood in a small test tube and will post back on the same day to a laboratory in London. Tests will be done twice: after the first and second vaccine doses.

The study will help us understand if the body's immune response to the COVID-19 vaccine is different in people with severe asthma who are on different treatments to manage their symptoms.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 16 years
2. For asthma patients:

   1. Diagnosis of severe asthma (based on ATS/ERS consensus criteria)
   2. Group A: Currently receiving an asthma biologic with treatment having started at least 3 months before first COVID-19 vaccine
   3. Group B: on maintenance oral steroids at a dose of ≥5mg prednisolone (or equivalent) per day (at the time of first COVID-19 vaccine)
   4. Group C: not on asthma biologic or maintenance oral steroids (at the time of vaccination) or stopped ≥3 months prior to first COVID-19 vaccine

Exclusion criteria:

1. Current pregnancy or planning a pregnancy within the next 6 months
2. Current malignancy
3. Diagnosis of immunodeficiency requiring treatment
4. Additional exclusion criteria for asthma patients:

   1. Group A: maintenance oral steroids at the time of first COVID-19 vaccine
   2. Group B: on an asthma biologic at the time of first COVID-19 vaccine
5. Additional exclusion criteria for healthy controls cohort (as assessed by research team):

   1. No history of asthma or significant other lung disease
   2. Severe chronic inflammatory disease
   3. Severe cardiac disease
   4. Diabetes
6. Previous proven COVID-19 infection
7. Inability to provide informed consent
8. Unwilling to have vaccination
9. Participation in another clinical trial involving an investigational medicinal product (IMP).

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit patients that attended the severe asthma clinic. To recruit age-matched controls we will randomly approach the patients and ask if their partners (or age-matched family members or friends) would like to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Measured immune response | 12 Months
  To compare the measured immune response to vaccination in patients with 200 severe asthma and 50 healthy individuals. A positive response will be defined as IgG ≥0.201.

SECONDARY OUTCOMES:
Range of immune responses | 12 Months
  To evaluate the range of immune responses measured by IgG titres (very high: >1.25, high: 0.751-1.25, medium: 0.401-0.75 or low: 0.201-0.4) in patients with 200 severe asthma and compare this with 50 healthy individuals
Differences in responses between treatment groups | 12 Months
  To identify any differences in responses between patients treated with biologics, standard inhaler treatment with/without maintenance oral corticosteroids (mOCS)
Differences between responses within the three biologics | 12 Months
  To identify any differences between responses to vaccines amongst patient groups treated with three biologics (anti-IgE Omalizumab, anti-IL-5 Mepolizumab, and anti-IL-5receptor Benralizumab)

CONTACTS AND LOCATIONS:
Overall Officials: Hitasha Rupani, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Gartnavel General Hospital, Glasgow
  - Guy's and St Thomas' NHS Trust Foundation, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cates CJ, Rowe BH. Vaccines for preventing influenza in people with asthma. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD000364. doi: 10.1002/14651858.CD000364.pub4. PMID 23450529